CLINICAL TRIAL: NCT03575338
Title: Minimally Invasive Versus Open Scarf Osteotomy for Hallux Valgus Correction: a Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Responsible Party: Principal Investigator, josep torrent, Josep Torrent m.d., Hospital Mutua de Terrassa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hospital Mútua Terrassa
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Hallux Valgus and Bunion (Disorder)
Keywords: scarf; minimally invasive surgery; hallux valgus
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will not know the technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Scarf Osteotomy (Active Comparator): This group of patients will undergo surgery performing an open scarf osteotomy
  Interventions: Procedure: Open Scarf Osteotomy
- Minimally invasive scarf Osteotomy (Experimental): This group of patients will undergo surgery performing a Minimally invasive scarf osteotomy
  Interventions: Procedure: Minimally invasive scarf Osteotomy

INTERVENTIONS:
Procedure: Open Scarf Osteotomy — Open Scarf Osteotomy
  Arms: Open Scarf Osteotomy
Procedure: Minimally invasive scarf Osteotomy — Minimally invasive scarf Osteotomy
  Arms: Minimally invasive scarf Osteotomy

SUMMARY:
The purpose of this study was to compare a minimally invasive scarf technique and the well-established open scarf technique for correction of hallux valgus deformity.

DETAILED DESCRIPTION:
Hallux valgus surgery is a common procedure being the open scarf osteotomy, one of the most studied techniques for correction of the hallux valgus. It is widely reported its capacity to reduce the angle of the first metatarso-phalangeal joint.

Minimally invasive scarf (MIS) technique has been designed to decrease the soft tissue damage and postoperative pain. This procedure does not require ischemia, being able to do under local anesthesia and sedation. This technique is more suitable for outpatient surgery.

There is a lack of studies comparing both techniques, and our purpose is to do a prospective comparative study among the two approaches of the scarf osteotomy: open vs MIS.

ELIGIBILITY:
Inclusion Criteria:

- Patients undergo hallux valgus surgery

Exclusion Criteria:

* Intermetatarsal angle >20º
* Previous hallux valgus surgery
* Metatarsalgia of the lesser rays that requires an osteotomy during the surgical procedure
* 1st cuneometatarsal instability
* Infection
* Vascular ischemia
* Neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Hallux valgus angle postoperative | 1 year - 2 years
  The angle among the first metatarsal and the first phalanx

SECONDARY OUTCOMES:
Intermetatarsal 1-2 angle | 1 year - 2 years
  The angle among the 1st and the 2nd metatarsal
First metatarso-phalangeal range of movement | 1 year - 2 years
  The range of movement of the first metatarso-phalangeal joint
Surgery duration | Measurement during the surgery
  The records of the surgery duration
Irradiation | Measurement during the surgery
  The records of the radiation during the surgeries

CONTACTS AND LOCATIONS:
Locations (1):
- Josep Torrent, Terrassa, Barcelona, Spain